CLINICAL TRIAL: NCT06887296
Title: Assessment of the Impact of Polycystic Ovary Syndrome on Women's Sexuality
Acronym: SexOPK
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0135; ID-RCB : 2025-A00613-46 (Other: ANSM)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
Keywords: Polycystic Ovary Syndrome; Female Sexuality; Quality of Life; Sexual Health
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with polycystic ovary syndrome
  Interventions: Other: women answer a questionnaire
- Women without polycystic ovary syndrome
  Interventions: Other: women answer a questionnaire

INTERVENTIONS:
Other: women answer a questionnaire — Sexual Function and Distress Assessment in Women with Polycystic Ovary Syndrome (PCOS) Using Standardized Questionnaires

SUMMARY:
This study, titled SexOPK, aims to evaluate the impact of polycystic ovary syndrome (PCOS) on women's sexual health. PCOS is a common endocrine disorder affecting 5-20% of women of reproductive age, often leading to hormonal imbalances, metabolic issues, and psychological distress. Despite existing studies on the subject, the level of sexual distress associated with PCOS-related sexual dysfunction remains unclear.

The study will compare sexual function and distress levels between women diagnosed with PCOS and a control group without PCOS. Participants will complete an online questionnaire assessing various aspects of sexual health, body image, anxiety, and depression. The findings may help healthcare professionals better understand and address sexual dysfunction in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

For patients in the test group (PCOS):

* Adults
* Carriers of medically diagnosed polycystic ovarian syndrome
* Non-opposition

For patients in the control group:

* Adults
* Not carriers of polycystic ovarian syndrome
* Unopposed

Exclusion Criteria:

* Patient under court protection, guardianship, or curatorship
* Does not understand or speak French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of women with or without polycystic ovary syndrome to constitute 2 groups of 40 participants.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of Sexual Function and Distress in Women with Polycystic Ovary Syndrome Using BISF-W Scores | Day 1
  The Brief Index of Sexual Functioning for Women (BISF-W) is a validated questionnaire that assesses various aspects of female sexual function, including desire, arousal, frequency of sexual activity, receptivity, orgasm, satisfaction, and concerns affecting sexuality. It consists of 22 items, generating a composite score that reflects overall sexual well-being. Higher BISF-W scores indicate better sexual function, while lower scores suggest sexual dysfunction or distress.
Evaluation of Sexual Function and Distress in Women with Polycystic Ovary Syndrome Using FSDS-R Scores | Day 1
  The Female Sexual Distress Scale-Revised (FSDS-R) is a 13-item questionnaire designed to measure sexual distress in women, including feelings of frustration, guilt, stress, and dissatisfaction related to sexual activity. The total score ranges from 0 to 52, with higher scores indicating greater sexual distress and lower scores reflecting better emotional well-being regarding sexuality

SECONDARY OUTCOMES:
Assessment of Body Image Satisfaction Using the QIC Questionnaire | Day 1
  The third part corresponds to the QIC questionnaire (Body Image Questionnaire), which includes 19 items and explores body satisfaction/dissatisfaction indirectly, by taking into account a set of desirable/undesirable bodily attributes and states
Evaluation of Anxiety and Depression Using the HADS Scale | Day 1
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire designed to assess anxiety and depression symptoms in non-psychiatric medical settings. It consists of two subscales: HADS-A (7 items for anxiety) and HADS-D (7 items for depression). Each item is scored from 0 to 3, leading to subscale scores ranging from 0 to 21 and a total score from 0 to 42.
  For each subscale, a lower score (0-7) indicates normal emotional status, 8-10 suggests a borderline case, and 11-21 reflects clinically significant anxiety or depression. A higher total score indicates greater psychological distress, while a lower score reflects better mental well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Gosset, Principal Investigator — University Hospital of Toulouse
Locations (1):
- CHU Paule de Viguier, Toulouse, France

IPD SHARING:
Plan to Share IPD: No